CLINICAL TRIAL: NCT01495195
Title: Combined Donepezil and Selegiline Effects on Cocaine-Reinforced Behavior
Acronym: SDC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Midwest Biomedical Research Foundation (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, KENNETH GRASING, Director, Substance Abuse Research Laboratory, Kansas City VA Medical Center, Midwest Biomedical Research Foundation
Organization: Midwest Veterans' Biomedical Research Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NCT01406522B; R21DA029787 (NIH)
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Cocaine Use Disorders
Keywords: Acetylcholine; Cholinesterases; Cocaine; Self-Administration
MeSH Terms: interventions — Donepezil; Selegiline

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Donepezil, high-dose (Experimental): Titration of donepezil to 22.5 mg daily
  Interventions: Drug: High-dose donepezil
- Selegiline & low-dose donepezil (Experimental): Low-Dose Donepezil [titrated to 10 mg daily] and transdermal selegiline [6 mg daily]
  Interventions: Drug: Low-dose donepezil; Drug: Selegiline
- Selegiline & high-dose donepezil (Experimental): High-Dose Donepezil [titrated to 22.5 mg daily] and transdermal selegiline [6 mg daily]
  Interventions: Drug: High-dose donepezil; Drug: Selegiline
- Sugar pill (Placebo Comparator): Inert pill for comparison
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: High-dose donepezil — Donepezil titrated to 22.5 mg daily
  Other Names: Aricept
  Arms: Donepezil, high-dose; Selegiline & high-dose donepezil
Drug: Low-dose donepezil — Donepezil titrated to 10 mg daily
  Other Names: Aricept
  Arms: Selegiline & low-dose donepezil
Drug: Selegiline — Transdermal selegiline, 6 mg daily
  Other Names: EMSAM
  Arms: Selegiline & high-dose donepezil; Selegiline & low-dose donepezil
Drug: Placebo — microcrystalline cellulose
  Arms: Sugar pill

SUMMARY:
No medications are currently available for treatment of psychostimulant addiction, a compulsive preoccupation with use of cocaine and related compounds. Donepezil is a medication that is currently prescribed for Alzheimer's disease, and selegiline is a medication used for treatment of Parkinson's Disease. Both of these medications can decrease the amount of cocaine injections that laboratory animals choose to inject by vein. This project will determine if combined treatment with donepezil and selegiline can also decrease cocaine-motivated behavior for human subjects in a laboratory setting.

DETAILED DESCRIPTION:
Background:

We have recently shown that pretreatment with certain cholinesterase inhibitors can produce large reductions in cocaine-reinforced behavior in rats (drug self-administration is decreased by more than 70% over a period of three days during which no additional cholinesterase inhibitor is administered). Because the reductions persist over a period two or more weeks, they have been described as persistent attenuation. Similar reductions have been observed after rats receive pretreatment with the cholinesterase inhibitors donepezil or tacrine, but not rivastigmine. The key difference leading to persistent attenuation may be effects of donepezil or tacrine on catecholamine neurotransmitters. Specifically, our hypothesis is that persistent attenuation is caused by a combination of 1.) Cholinesterase inhibition, which increases brain levels of acetylcholine (ACh); and 2.) Increased brain levels of dopamine and serotonin. Although well-tolerated, pretreatment with low doses of the cholinesterase inhibitor donepezil have not modified either the positive subjective effects of cocaine in humans, or cocaine use in outpatients. This may reflect the relatively low doses of donepezil administered (up to 10 mg daily). Transdermal selegiline is a well-tolerated, nonselective monoamine oxidase inhibitor that potentiates actions of dopamine and serotonin in the central nervous system.

Rationale Persistent attenuation may be achieved in humans by administering donepezil at higher doses, or in combination with a centrally-acting inhibitor of monoamine oxidase (MAO). Inhibition of MAO increases brain levels of dopamine and serotonin. If persistent attenuation can be accomplished in humans, this would lead to an important paradigm shift for substance abuse treatment, in that large reductions in cocaine-reinforced behavior could be produced without the need for continuous dosing with a medication. This scenario could remove the requirement for continued compliance with oral dosing in some patients with its associated potential for toxicity.

Specific Aims:

1. Determine whether donepezil can be safely advanced over a 17-day period to an individualized dose of up to 22.5 mg daily (or the highest dose tolerated by each participant).
2. Evaluate whether high-dose donepezil attenuates cocaine-reinforced behavior in humans.
3. Determine whether combined donepezil and selegiline produces greater reductions in cocaine-reinforced behavior than observed for donepezil alone.

Methods This is a randomized, single-blind, placebo-controlled, research-unit, single-center evaluation of the potential for oral donepezil, with or without transdermal selegiline to modify cocaine self-administration in a laboratory setting. Up to 32 non-treatment-seeking, regular cocaine users will be assigned to receive one of four treatments: 1.) Oral placebo; 2.) High-Dose Donepezil [titrated to 22.5 mg daily]; and 3.) Low-Dose Donepezil [titrated to 10 mg daily] and transdermal selegiline [6 mg daily]; and 4.) High-Dose Donepezil [titrated to 22.5 mg daily] and transdermal selegiline [6 mg daily]. For participants who receive donepezil, it will be advanced to either a target dose (low or high), or a lower dose that is tolerated by individual participants. To evaluate the occurrence of persistent attenuation, cocaine use will be measured over a nine-day follow-up period, through urine drug screens and the timeline-follow-back method. As noncontingent infusions of cocaine are administered, the pharmacokinetics of cocaine and donepezil will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV-TR criteria for cocaine abuse or dependence
* At least one cocaine-positive urine within 6 weeks prior to enrollment
* Has used cocaine for a duration of at least 6 months
* At least weekly cocaine use during the last 30 days

Exclusion Criteria:

* History of a medical adverse reaction to cocaine or other psychostimulants
* Any current Axis I psychiatric disorder other than drug abuse or dependence
* Dependence on abused substances other than cocaine
* Current or past history of seizure disorder
* Heart or lung disease

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Changes in cocaine-reinforced behavior | days 2 and 24 of dosing
  Participants will make a series of choices between vouchers with an ascending monetary value and intravenous injections of cocaine

SECONDARY OUTCOMES:
How well the study medications are tolerated | 33 days of dosing
  Laboratory and self-reported adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Kansas City VA Medical Center, Kansas City, Missouri, United States

REFERENCES:
- [Background] Grasing K, Mathur D, Newton TF, DeSouza C. Donepezil treatment and the subjective effects of intravenous cocaine in dependent individuals. Drug Alcohol Depend. 2010 Feb 1;107(1):69-75. doi: 10.1016/j.drugalcdep.2009.09.010. PMID 19836169
- [Background] Grasing K, Yang Y, He S. Reversible and persistent decreases in cocaine self-administration after cholinesterase inhibition: different effects of donepezil and rivastigmine. Behav Pharmacol. 2011 Feb;22(1):58-70. doi: 10.1097/FBP.0b013e3283428cd8. PMID 22173266